CLINICAL TRIAL: NCT00831129
Title: Effects of Simvastatin and Rosiglitazone Combination in Patients With the Metabolic Syndrome.
Brief Title: A Study for Pre-diabetic Patients With Cholesterol Lowering Drugs
Acronym: SIROCO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 14863B (SIROCO)
Record Dates: First submitted 2009-01-26; First posted 2009-01-28 (Estimated); Results first posted 2013-09-12 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Pre-diabetes
MeSH Terms: conditions — Glucose Intolerance | interventions — Rosiglitazone; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simvastatin + Placebo Rosiglitazone (Active Comparator): Subjects will receive 40 mg Simvastatin + 1 tab Placebo Rosiglitazone daily
  Interventions: Drug: Placebo Rosiglitazone; Drug: Simvastatin
- Simvastatin + rosiglitazone (Active Comparator): Subjects will receive 40 mg Simvastatin + 4 mg Rosiglitazone once daily
  Interventions: Drug: Rosiglitazone; Drug: Simvastatin

INTERVENTIONS:
Drug: Rosiglitazone — 4 mg daily
  Other Names: Avandia
  Arms: Simvastatin + rosiglitazone
Drug: Placebo Rosiglitazone — 1 tab daily
  Other Names: Placebo
  Arms: Simvastatin + Placebo Rosiglitazone
Drug: Simvastatin — 40 mg daily
  Other Names: Zocor

SUMMARY:
The purpose of this research study is to examine if a combination of a cholesterol lowering-drug, simvastatin, with a sugar-lowering drug called rosiglitazone is more effective in improving vascular inflammation (irritation of the vessels that transport your blood) and other cardiovascular risk factors than the taking of simvastatin alone.

DETAILED DESCRIPTION:
Age 21-75 years Metabolic syndrome (must have 3 of the 5 components) elevated waist circumference >40inches in men, >35 inches in women elevated triglycerides >150mg/dL reduced HDL <40mg/dL in men<50 in women elevated blood pressure >130mmHg systolic, or >85mmHg diastolic elevated fasting glucose >100mg/dL

ELIGIBILITY:
Inclusion Criteria:

* 21-75 years
* Metabolic syndrome (3 of the 5 components)
* Elevated waist circumference >40inches in men, >35inches in women
* Elevated triglycerides >150mg/dL
* Reduced HDL <40mg/dL in men, <50mg/dL in women
* Elevated blood pressure >130mmHg systolic, >85mmHg diastolic
* Elevated fasting glucose >100mg/dL

Exclusion Criteria:

* Diabetes mellitus
* Stage 3 hypertension >180mmHg systolic, >110mmHg diastolic office blood pressure
* History of non-diabetic kidney disease
* Myocardial infarction of unstable angina within the past 6 months
* History of liver disease
* History of malignancy
* History of drug or alcohol abuse
* Treatment with corticosteroids
* Pregnancy or lactating women of women of child bearing potential who are not willing to use reliable contraception method during the study

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2006-09; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Bakris, M.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: simvastatin 40 mg/day plus placebo
- Rosiglitazone: simvastatin 40 mg/day plus rosiglitazone 4 mg/day
Period: Overall Study
Arm/Group | Placebo | Rosiglitazone
Started | 20 | 33
Completed | 20 | 23
Not Completed | 0 | 10
Not completed — Adverse Event | 0 | 1
Not completed — 9 lost to follow-up reasons uknown | 0 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rosiglitazone | Total
Number analyzed (Participants) | 20 | 23 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (9.3) | 58.7 (12.1) | 57.03 (10.7)
Gender [Count of Participants; unit: Participants]
  Female | 6 | 14 | 20
  Male | 14 | 9 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change in High-sensitivity C-reactive Protein
Description: change in high-sensitivity C-reactive between baseline and 6 month
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 20 | 23
mg/dl | 0.72 (2.49) | -0.61 (1.36)

2. Secondary Outcome: Change in Urinary Isoprostane
Description: change in urinary isoprostane between baseline and 6 month
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 20 | 23
ng/ml | -0.79 (2.1) | -1.09 (1.9)

3. Secondary Outcome: Change in Malondialdehyde
Description: change in Malondialdehyde between baseline and 6 month
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 20 | 23
nM | -1.27 (2.4) | -1.52 (3.0)

4. Secondary Outcome: Change in Office Systolic Blood Pressure
Description: change in office systolic blood pressure between baseline and 6 month
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 20 | 23
mm Hg | -18.24 (12.5) | -16.77 (15.2)

5. Secondary Outcome: Change in Office Diastolic Blood Pressure
Description: change in office diastolic blood pressure between baseline and 6 month
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 20 | 23
mm Hg | -9.59 (9.9) | -9.46 (8.4)

6. Secondary Outcome: Change in (Ambulatory Blood Pressure Monitoring) Systolic Blood Pressure
Description: change in (ambulatory blood pressure monitoring) systolic blood pressure between baseline and 6 month
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 20 | 23
mm Hg | 3.41 (3.7) | -1.08 (1.2)

7. Secondary Outcome: Change in (Ambulatory Blood Pressure Monitoring) Diastolic Blood Pressure
Description: change in (ambulatory blood pressure monitoring) diastolic blood pressure between baseline and 6 month
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 20 | 23
mm Hg | -0.88 (0.9) | -0.69 (0.6)

8. Secondary Outcome: Change in Low-density Lipoprotein
Description: change in low-density lipoprotein between baseline and 6 month
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 20 | 23
mg/dl | -38.88 (41.2) | -28.77 (31.7)

9. Secondary Outcome: Change in Triglycerides
Description: change in Triglycerides between baseline and 6 month
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 20 | 23
mg/dl | -34.32 (22.1) | -42.47 (27.3)

10. Secondary Outcome: Change in High-density Lipoprotein
Description: change in high-density lipoprotein between baseline and 6 month
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 20 | 23
mg/dl | 0.71 (7.9) | 2.77 (6.7)

11. Secondary Outcome: Change in Glycosylated Haemoglobin
Description: change in glycosylated haemoglobin between baseline and 6 month
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 20 | 23
percentage of glycosylated haemoglobin | 0.12 (0.11) | -0.22 (0.07)

12. Secondary Outcome: Change in Fasting Blood Glucose
Description: change in fasting blood glucose between baseline and 6 month
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 20 | 23
mg/dl | 5.94 (10.9) | -4.85 (11.3)

13. Secondary Outcome: Change in Insulin
Description: change in Insulin between baseline and 6 month
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: IU/ml
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 20 | 23
IU/ml | 0.59 (1.1) | -3.47 (1.8)

14. Secondary Outcome: Change in Homeostatic Model Assessment for Insulin Resistance
Description: change in homeostatic model assessment for insulin resistance between baseline and 6 month
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: HOMA units
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 20 | 23
HOMA units | 0.31 (1.4) | -2.08 (2.8)

15. Secondary Outcome: Change in Adiponectin
Description: change in Adiponectin between baseline and 6 month
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: μg/ml
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 20 | 23
μg/ml | -0.24 (1.3) | 4.15 (3.9)

16. Secondary Outcome: Change in Body Mass Index
Description: change in body mass index between baseline and 6 month
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Placebo | Rosiglitazone
Number analyzed (Participants) | 20 | 23
kg/m2 | -0.21 (2.18) | 0.68 (1.1)

ADVERSE EVENTS:
Arm/Group | Placebo | Rosiglitazone
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/23
Other Adverse Events (participants affected / at risk) | 6/20 | 9/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | Rosiglitazone (N=23)
Nonspecific muscle aches in lower extremities (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Nausea Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper respiratory symptoms (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Headaches (Nervous system disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Joint aches (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) — vague complaints of joint aches involving the knee, hip or ankle in all cases at least 2 or more of these joints

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes